CLINICAL TRIAL: NCT03810898
Title: First-in-Human Adaptive Study to Investigate the Binding and Kinetic Properties of Two Novel PET Ligands and Their Suitability for Quantification of Aggregated Mutant Huntingtin in the Brains of Huntington's Disease Gene-Expansion Carriers
Brief Title: iMagemHTT: FIH Evaluation of Novel Mutant Huntingtin PET Radioligands [¹¹C]CHDI-00485180-R and [¹¹C]CHDI-00485626
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study terminated per protocol design post interim analysis review after Phase 2a. No SAEs or safety issues were noted.
Sponsor: CHDI Foundation, Inc. (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: C-000418-2
Record Dates: First submitted 2018-12-07; First posted 2019-01-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; Huntington's Disease; HD; HDGEC; Gene Expansion Carrier; PET; Tracer; Positron Emission Tomography; radioligand; imaging; mHTT; huntingtin; iMagemHTT
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: Huntington's disease gene expansion carriers (HDGEC) compared to healthy controls (HC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1 (a & b) (Experimental): Radioligand [¹¹C]CHDI-00485180-R and/or Radioligand [¹¹C]CHDI-00485626/ 6 Stage II HDGECs and 6 young (< 35) HCs/ Imaging- MRI and PET/
  Both radioligands administered- 1x each/ Optional CSF collection for HDGECs
  Interventions: Radiation: Radioligand [¹¹C]CHDI-00485180-R; Radiation: Radioligand [¹¹C]CHDI-00485626
- Phase 2a (Experimental): Per Radioligand- Radioligand [¹¹C]CHDI-00485180-R or Radioligand [¹¹C]CHDI-00485626/ 6 Stage II HDGECs and 6 age matched HCs/ Imaging- MRI and PET/
  1 Radioligand administered 2x (test re-test)- HDGECs/ Optional CSF collection for HDGECs
  1 Radioligand administered 1x- HCs/
  Interventions: Radiation: Radioligand [¹¹C]CHDI-00485180-R; Radiation: Radioligand [¹¹C]CHDI-00485626
- Phase 2b (Experimental): Per Radioligand- Radioligand [¹¹C]CHDI-00485180-R or Radioligand [¹¹C]CHDI-00485626/ 6 Stage I HDGECs and 6 age matched HCs/ Imaging- MRI and PET/
  1 Radioligand 1 or 2x administered (test re-test optional)- HDGECs/ Optional CSF collection for HDGECs
  1 Radioligand administered 1x -HCs/
  Interventions: Radiation: Radioligand [¹¹C]CHDI-00485180-R; Radiation: Radioligand [¹¹C]CHDI-00485626
- Phase 2c (Experimental): Per Radioligand- Radioligand [¹¹C]CHDI-00485180-R or Radioligand [¹¹C]CHDI-00485626/ 6 Pre-manifest HDGECs and 6 age matched HCs/ Imaging- MRI and PET/
  1 Radioligand administered 1 or 2x (test re-test optional)- HDGECs/ Optional CSF collection for HDGECs
  1 Radioligand administered 1x- HCs/
  Interventions: Radiation: Radioligand [¹¹C]CHDI-00485180-R; Radiation: Radioligand [¹¹C]CHDI-00485626

INTERVENTIONS:
Radiation: Radioligand [¹¹C]CHDI-00485180-R — Intravenous injection of radioligand in the arm with PET imaging of the brain.
Radiation: Radioligand [¹¹C]CHDI-00485626 — Intravenous injection of radioligand in the arm with PET imaging of the brain.

SUMMARY:
This is a FIH (first-in-human) adaptive PET (Positron Emission Tomography) imaging study to explore the binding and kinetic properties of two potential mutant huntingtin (mHTT) radioligands; [¹¹C]CHDI-00485180-R and [¹¹C]CHDI-00485626.

The binding characteristics of these radioligands will be evaluated first in young (< 35 years of age) healthy control (HC) participants (Phase 1a) and subsequently in young HCs and Huntington's disease gene-expansion carriers (HDGECs) with Stage II HD (Phase 1b). Subsequent phases will continue to explore the radioligands' binding characteristics in HDGECs with Stage II HD (Phase 2a), Stage I HD (Phase 2b) and pre-manifest HDGECs (Phase 2c) and their age matched healthy controls. All phases are cross-sectional and will include comparisons between HCs and HDGECs. Test-retest (TRT) evaluations will be done during Phase 2a, with the option of including further test-retests in Phases 2b, and 2c after review of data by the iMagemHTT Executive Committee. TRT is only applicable to HDGEC participants.

There are four planned interim analyses at which either radioligand may be dropped if its characteristics are shown to be suboptimal. If successful, the study will establish [¹¹C]CHDI-00485180-R and/or [¹¹C]CHDI-00485626 as fit for further development as drug development tools to measure mHTT levels in HDGECs. This development is intended to demonstrate the value of PET imaging with these radioligands as a disease progression biomarker, predictive biomarker, pharmacodynamic biomarker, and eventually as an efficacy biomarker.

All HDGEC participants will be invited to provide an optional cerebrospinal fluid (CSF) sample that will be collected after the imaging visits are complete. These samples will be processed to evaluate CSF mHTT levels and other potential biomarkers and to explore potential relationships between soluble CSF mHTT levels and mHTT binding identified by [¹¹C]CHDI-00485180-R and/or [¹¹C]CHDI-00485626 PET imaging. Potential CSF biomarkers that might be co-expressed or accumulated in HD may also be examined.

DETAILED DESCRIPTION:
The study investigators have developed two novel PET radioligands that will be evaluated for their suitability for use in clinical research settings to quantify mHTT in HDGECs. The PET radioligands do not have any pharmacological effect at the microdoses (total dose <100ug) at which they will be administered; they will not be administered at pharmacological doses. This study has a modular design in two phases, and each phase will enroll a small independent cohort. The execution of each subsequent phase is dependent on results from the previous phase.

Phase 1 is the initial evaluation of the PET radioligands. A suitable PET radioligand is expected to produce quantifiably higher binding in HD participants' brains compared to young HC participants' brains (since they do not express mHTT). Phase 1 is divided in two sub phases: Phase 1a will evaluate the basic safety and kinetic properties as well as brain uptake in three (3) young HCs; Phase 1b will test the difference in binding in six (6) HDGECs with Stage II HD compared to six (6) young HCs (three (3) young HCs will be imaged in addition to the three (3) young HCs from 1a. The rationale behind using young HCs in Phase 1 is to screen out HC participants who may have undiagnosed amyloid-β (Aβ) plaques, a potential off-target binding site for [¹¹C]CHDI-00485180-R. The rationale behind imaging HDGECs with Stage II HD in Phase 1 is based on the hypothesis that the density of mHTT aggregates increases with disease severity, and the ability to detect a difference in binding between HCs and HDGECs is expected to be higher in Stage II HD (more severe stages of HD will not be included in this study). An option to image three (3) pre-manifest HDGECs from Phase 2c (see below) will be included in case the results indicate that brain atrophy (i.e., loss of aggregate due to atrophy) affects the binding and evaluation of the PET radioligands in HDGECs with Stage II HD. For each of the two PET radioligands a Go/ No-Go evaluation will take place (for overview see Figure 1); if satisfactory results are not obtained for a particular radioligand, then that radioligand will not progress to evaluation in further phases. Promising results for either radioligand will lead to that particular radioligand continuing to Phase 2 evaluation.

Phase 2 will evaluate the sensitivity of the PET radioligand(s) to discriminate between different stages and severity of HD. In addition, a TRT in Phase 2 will evaluate the variability of repeated imaging for the PET radioligand. Phase 2 has a sequential design in sub phases that will assess the sensitivity of the radioligand in descending severity of HD: 2a in six (6) HDGECs with Stage II HD and six (6) age-matched controls; 2b in six (6) HDGECs with Stage I HD and six (6) age-matched controls; 2c in six (6) premanifest HDGECs and six (6) age-matched controls. The rationale for imaging groups of descending HD severity is based on the hypothesis that the density of mHTT aggregates increases with disease severity, and the ability to detect a difference in binding between HCs and HDGECs is expected to be lowest in the premanifest stage. This design will enable a stepwise assessment of the sensitivity of the PET radioligands. After each sub-phase a Go/No-Go evaluation will take place; if satisfactory results are not obtained for a particular radioligand then that radioligand will not be evaluated in further sub-phases. Promising results for either radioligand will lead to that particular radioligand continuing to the next sub-phase.

This study design allows each radioligand to be reviewed and analyzed after evaluation in each cohort. The progression through each level of analysis will indicate whether either or both radioligands will measure mHTT aggregate levels with sufficient sensitivity to become potential disease progression and efficacy biomarker(s) in HDGECs.

ELIGIBILITY:
Inclusion Criteria:

Pre-manifest HDGECs, HDGECs with Stage I HD, HDGECs with Stage II HD and HC participants:

* Female and male adults, age 20-65 years old, inclusive.
* Body Mass Index (BMI) between 19 and 35 inclusive.
* Capacity to give full informed consent in writing, and have read and signed the informed consent form (ICF).
* Are capable of complying with study procedures, including fasting and blood sampling
* Able and willing to travel to imaging PET center in Leuven, Belgium.
* Willing to comply with the use of adequate contraceptive measures.

Pre-manifest HDGECs:

* Do not have clinical diagnostic motor features of HD, defined as Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Score < 4; and
* Have CAG expansion ≥ 40; and
* Have a CAP score > 70 (as calculated with CAP formula: AGE * (CAG - 30) / 6.49).

HDGECs with Stage I HD:

* Have clinical diagnostic motor features of HD, defined as UHDRS Diagnostic Confidence Score = 4; and
* Have CAG expansion ≥ 40; and
* Have Stage I HD, defined as UHDRS Total Functional Capacity (TFC) scores between 11 and 13 inclusive.

HDGECs with Stage II HD:

* Have clinical diagnostic motor features of HD, defined as UHDRS Diagnostic Confidence Score = 4; and
* Have CAG expansion ≥ 40; and Have Stage II HD, defined as UHDRS Total Functional Capacity (TFC) scores between 7 and 10 inclusive.

HC participants:

* Have no known family history of HD; or
* Have known family history of HD but have been tested for the huntingtin gene glutamine codon (CAG) expansion and are not at genetic risk for HD (CAG < 36).
* Matched by age +/- 5 years.
* (Phase 1 only) under 35 years of age.

Exclusion Criteria:

Pre-manifest HDGECs, HDGECs with Stage I HD, HDGECs with Stage II HD, and HC participants:

* Currently participating in or less than 30 days after completing participation in other therapeutic or imaging studies.
* Previous participation in PET imaging study that, cumulatively with the current study, will exceed annual regulatory limits for radiation exposure.
* Any disease, condition, or concomitant medication that significantly compromises the function of the body systems and that in the opinion of the Investigator, might interfere with the conduct of the study or its interpretation.
* Pregnant and breastfeeding females.
* Concomitant medication (ConMed) use of antiplatelet or anticoagulant therapy (inclusive of acetylsalicylic acid). (See full ConMed list attached.)
* Needle phobia.

HDGEC participants:

• If using any antidepressant, psychoactive, psychotropic or other medications or nutraceuticals used to treat HD, the use of inappropriate (e.g., non-therapeutically high) or unstable dose within 30 days prior to participation.

HC participants:.

• Family history of HD (unless genetic test confirming negative results).

For participants in optional CSF sample collection:

* Frequent headache, significant lower spinal deformity or major surgery; or
* Bleeding disorder.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
The VT (volume of distribution total) of 2 discrete PET markers will be measured with PET imaging. | Single point measure- 90 minutes scan
  VT (volume of distribution total) is derived from the data collected during each PET scan. VT is the amount of the PET marker in a volume of tissue (i.e., a concentration).

CONTACTS AND LOCATIONS:
Overall Officials: Wim Vandenberghe, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen Leuven/ UZ Leuven/ UZL; Mette Skinbjerg, PhD, Study Director — CHDI Management/ CHDI Foundation
Locations (1):
- Universitaire Ziekenhuizen Leuven/ UZ Leuven/ UZL, Leuven, Belgium

REFERENCES:
- [Derived] Delva A, Koole M, Serdons K, Bormans G, Skinbjerg M, Khetarpal V, Liu L, Bard J, Doot R, Warner JH, Sathe S, Sampaio C, Wood A, Van Laere K, Vandenberghe W. PET imaging with [(1)(1)C]CHDI-00485180-R, designed as radioligand for aggregated mutant huntingtin, in people with Huntington's disease. Eur J Nucl Med Mol Imaging. 2025 Nov;52(13):5124-5134. doi: 10.1007/s00259-025-07394-w. Epub 2025 Jun 18. PMID 40527969